CLINICAL TRIAL: NCT00367406
Title: Comparison Between Gamma 3 Nail and ACE Trochanteric Nail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/280
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2014-12

CONDITIONS: Pertrochanteric and Subtrochanteric Femur Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with a Gamma 3 nail. (Experimental)
  Interventions: Device: Gamma 3 nail versus ACE trochanteric nail

INTERVENTIONS:
Device: Gamma 3 nail versus ACE trochanteric nail — Comparing Gamma 3 nail versus ACE trochanteric nail

SUMMARY:
Pertrochanteric and subtrochanteric femur fractures will be treated with a Gamma 3 nail or an ACE Trochanteric nail.

Following topics will be assessed: fracture consolidation, mobility, pain, walking power, agility.

ELIGIBILITY:
Inclusion Criteria:

* Pertrochanteric or subtrochanteric femur fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Consolidation of the fracture | From surgery untill healing

CONTACTS AND LOCATIONS:
Overall Officials: René Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be